CLINICAL TRIAL: NCT00045175
Title: A Phase I Study of UCN-01 in Combination With Topotecan in Patients With Solid Tumors
Brief Title: UCN-01 and Topotecan in Treating Patients With Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-005; CDR0000256917 (Registry Identifier: PDQ (Physician Data Query)); NCI-5518
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: primary peritoneal cavity cancer; recurrent ovarian epithelial cancer; fallopian tube cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — 7-hydroxystaurosporine; Topotecan

ARMS (1):
- UCN-01 in combination with topotecan (Experimental)
  Interventions: Drug: 7-hydroxystaurosporine; Drug: topotecan hydrochloride

INTERVENTIONS:
Drug: 7-hydroxystaurosporine
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Topotecan may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining chemotherapy with topotecan may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining UCN-01 with topotecan in treating patients who have recurrent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of UCN-01 and topotecan in patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the relationship between clinical and pharmacokinetic effects of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive UCN-01 IV over 3 hours on day 1 and topotecan IV over 30 minutes on days 1-5. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of UCN-01 and topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Up to 12 additional ovarian epithelial cancer patients are then treated at the recommended phase II dose.

Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 3-30 patients will be accrued for this study within 6-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer
* Measurable disease outside of field of prior radiotherapy OR
* Progressive disease within field after radiotherapy
* Must have had no more than 2 prior chemotherapy regimens

  * At least 1 prior regimen must have included a platinum agent (e.g., carboplatin or cisplatin)
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine no greater than ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular

* No coronary artery disease
* No symptomatic cardiac dysfunction
* No symptoms suggestive of coronary artery disease with evidence of cardiac pathology

Pulmonary

* No symptomatic pulmonary dysfunction

Other

* No prior allergic reaction attributed to compounds of similar chemical or biologic composition to UCN-01 or other agents used in this study
* No insulin-dependent diabetes mellitus
* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior biologic therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No prior topotecan (other prior topoisomerase I inhibitors allowed)

Endocrine therapy

* At least 4 weeks since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 40% of bone marrow
* No prior mediastinal irradiation

Surgery

* At least 4 weeks since prior surgery

Other

* Recovered from all prior therapy
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent combination antiretroviral therapy for HIV-positive patients

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-06; Primary Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal W. Hirte, MD, FRCP(C), Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (3):
- Canada (3):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario